CLINICAL TRIAL: NCT07320807
Title: The Effect of Extracorporeal Shock Wave Therapy on Range of Motion, Pain, Dexterity, and Function After Hand Flexor Tendon Injury.
Brief Title: Effects of Extracorporeal Shock Wave Therapy After Flexor Tendon Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Nazife Kapan, Asist.Prof., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AYBU-ESWT-MK-01
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Tendon Injury - Hand
Keywords: rehabilitation; ekstrakorporeal shock wave therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): In accordance with the Modified Duran Protocol, a hand rehabilitation program, including early passive mobilization, will be implemented for 4 weeks.
- intervention (Experimental): In addition to a hand rehabilitation program that includes early passive mobilization in accordance with the Modified Duran Protocol, ESWT will be applied.
  Interventions: Device: Ekstracorporeal Shock Wave Therapy

INTERVENTIONS:
Device: Ekstracorporeal Shock Wave Therapy — Radial ESWT with 2 bar pressure, 10 Hz frequency, and 2000 pulses will be applied to the flexor tendon scar tissue in a total of 4 sessions, once a week, using a sweeping method with gel applied between the patient's skin and the probe.
  Arms: intervention

SUMMARY:
In this study aims to investigate the effects of extracorporeal shock wave therapy, applied to the intervention group in addition to the rehabilitation program applied to the control and intervention groups, on range of motion, pain, grip strength, and dexterity after hand flexor tendon injury.

DETAILED DESCRIPTION:
The hand is a fundamental element in daily living activities, occupation, and social independence. Although different studies report varying figures for hand injuries, they constitute approximately 20% of injuries presenting to emergency departments. Soft tissue traumas account for a significant portion of these injuries. Due to the proximity of flexor tendons to the skin, the hand is frequently affected in hand injuries.

One of the agents used to accelerate healing and function in hand tendons after injury or surgery, and to reduce adhesion and contracture formation, is Extracorporeal Shock Wave Therapy (ESWT). ESWT treatment modalities have been tested in experimental animal studies. The idea behind the use of shock waves in the treatment of orthopedic diseases is to stimulate healing in tendons, surrounding tissues, and bones. The importance of shock wave therapy on soft tissues has increased over time.

It has been reported that ESWT significantly reduces deformity in Dupuytren's disease treatment. Brunelli et al. found that radial ESWT (3 bars, 12 Hz, 1400 pulses) applied in 4 sessions to a patient with pain, weakness in the middle and ring fingers, and flexion deformity due to Dupuytren's disease resulted in a significant reduction in hand deformities and improvement in daily living performance. Positive results of the use of ESWT in hand flexor tendon pathologies have been published. In their cadaver study examining the applicability of radial ESWT to the flexor tendon, Lutter et al. stated that ESWT application at different intensities can penetrate soft tissues and is a treatment option in different finger pathologies. Malliaropoulos et al. have found that radial ESWT is effective in reducing pain and improving functional recovery in trigger finger treatment. This study aims to investigate the effect of ESWT on range of motion, pain, grip strength, and dexterity after hand flexor tendon injury. 56 patients who presented with flexor tendon injury and consented to participate will be included in this study and divided into two groups. All patients will be enrolled in a hand rehabilitation program including early passive mobilization according to the Modified Duran Protocol. In addition, the intervention group will receive 2000 pulses of radial ESWT at 2 bar pressure and 10 Hz frequency, applied to the flexor tendon scar tissue in 4 sessions, using a sweeping method with gel applied between the patient's skin and the probe.

ELIGIBILITY:
Inclusion Criteria:

* • . Volunteering

  * . Being 8-12 weeks post-operatively after flexor tendon repair
  * . Having undergone flexor tendon zone II-IV surgical repair

Exclusion Criteria:

* . Infection

  * • . Open wound

    * . Pregnancy
    * . History of finger or wrist fracture
    * . Inflammatory rheumatic disease
    * . Malignant tumor mass

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Evaluation will be performed before treatment, on the day treatment ends, and one month after treatment.
  For VAS assessment, patients are informed about the meaning of the numbers placed on a 10 cm line from 0 to 10. It is explained that no pain is worth 0 points, moderate pain is worth 5 points, and the most severe pain felt is worth 10 points. Based on these explanations, the patient is asked to mark the pain on the 10 cm line. The distance between the marked point and the starting point is measured with a ruler to determine the pain intensity.
Range of Motion | Evaluation will be performed before treatment, on the day treatment ends, and one month after treatment.
  Range of motion (ROM) is one of the most frequently used outcome variables after tendon injuries in the hand. ROM measurement in the hand is performed using a finger goniometer. In active ROM assessment for the fingers, the patient is asked to make a fist for flexion and extend the finger straight; that is, the measurement is performed in a compound manner. In this study, the Modified Strickland calculation will be used for fingers 2-5. Active distal interphalangeal (DIF) and proximal interphalangeal (PIF) joint flexion are added together, and the active extension loss is subtracted. 175° is considered ideal and compared to 175°. The results are; 75°-100° is considered excellent, 50°-74° good, 25°-49° average, and 0°-24° poor.

SECONDARY OUTCOMES:
Nine-hole peg test | Evaluation will be performed before treatment, on the day treatment ends, and one month after treatment.
  Due to its low cost, ease of application, and speed, it is widely used in assessing dexterity. It consists of a square wooden board with nine holes and nine wooden pegs designed to fit these holes. During the test, the container with the square board and pegs is placed on the side of the extremity being evaluated. Then, the patient is asked to take the pegs one by one and place them in the holes. The order of placement is not important. As soon as the placement is complete, the pegs are removed one by one and returned to the container. The order of removal is not important. The process is timed. The timer starts when the hand first touches a peg at the beginning of placement and ends when the last peg is removed and touches the container.
Duruoz Hand Index | Evaluation will be performed before treatment, on the day treatment ends, and one month after treatment.
  The Duruoz Hand Index was first developed in 1996 to assess hand-related activity limitations in patients with Rheumatoid Arthritis. It consists of 18 self-assessed items regarding hand abilities in the kitchen, dressing, personal hygiene, work, and other general movements. Scores range from 0-40 for kitchen tasks, 0-10 for dressing, hygiene, and office tasks, and 0-20 for the "other" category. Individuals rate their abilities on a scale of 0 (no difficulty) to 5 (impossible to perform). The questionnaire results in a total score of 0-90. A higher score represents a greater activity limitation and greater difficulty. The validity and reliability of the Turkish version of the questionnaire have been demonstrated in patients with traumatic hand injuries.
Short Form-36 Questionnaire | Evaluation will be performed before treatment, on the day treatment ends, and one month after treatment.
  The Short Form-36 (SF-36) questionnaire is a 36-item scale consisting of subscales of physical function, physical role, emotional role, pain, vitality, general health, and mental health. Each subscale is scored from "0" to "100", indicating the lowest and highest quality of life levels, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No